CLINICAL TRIAL: NCT05452395
Title: Integrated Post-Acute Care Program for Frail Elderly
Brief Title: Post-acute Care for Patients With Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Tai-Yin Wu, Doctor, Taipei City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPECH-frailty
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Frailty; Retrospective Study
MeSH Terms: conditions — Frailty | interventions — Subacute Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-acute care (Experimental): comprehensive geriatric assessment, and either home-based or hospital-based post-acute care
  Interventions: Other: Post-acute care
- control group (No Intervention): comprehensive geriatric assessment only

INTERVENTIONS:
Other: Post-acute care — A personalized care program, focusing on managing geriatric syndromes and improving functional performances.
  Strength training, activities of daily living (ADL) and instrumental activities of daily living (IADL) practice, basic mobility training, reconditioning exercise, and home environment assessment and modification.
  Arms: Post-acute care

SUMMARY:
Acute illness could be enormous stress for frail people. Combining comprehensive geriatric assessment and multifactorial intervention has positive effects on frail community older adults. However, few studies investigated the effects of post-acute care (PAC) in frail older patients who just recovered from acute hospitalization. This study aimed to evaluate the effects of PAC on frail older adults in Taiwan.

DETAILED DESCRIPTION:
Frail patients aged >= 75 were recruited and divided into PAC or control groups. The PAC group received comprehensive geriatric assessment (CGA) and multifactorial intervention for two to four weeks. The control group received CGA only. The primary outcomes were 90-day emergency room visits, readmissions, and mortality after PAC.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to severe frailty identified by the Clinical Frailty Scale
2. Age ≥ 75 years
3. Diagnosis with Parkinson's disease, dementia, chronic obstructive pulmonary disease, or chronic kidney disease stage three or worse
4. Acute hospital stays between 3 to 30 days with deconditioning
5. Stable medical condition with no need of intensive care, laboratory examination, or oxygen dependence

Exclusion Criteria:

1. Refused to participate in the program
2. Candidate for other post-acute care programs (i.e. stroke, traumatic neurological injury, or fracture)
3. Unable to cooperate with the program due to mental or cognitive impairment
4. Long-term ventilator-dependence
5. Long-term bed-ridden status (> 6 months)
6. Diagnosed as end of life and in need of palliative care
7. Diagnosed as major illness (i.e. end-stage renal disease) and in need of frequent inpatient treatment ( > 3 times over recent 6 months)
8. Institutional residents
9. Home medical care participants

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 254 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
90-day emergency room visits | 90 days after post-acute care
  Emergency room visits after post-acute care
90-day readmissions | 90 days after post-acute care
  Readmissions visits after post-acute care
90-day mortality | 90 days after post-acute care
  Mortality after post-acute care

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Yin Wu, PhD, Principal Investigator — Department of Family Medicine, Taipei City Hospital, Zhongxing Branch
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lee MC, Wu TY, Huang SJ, Chen YM, Hsiao SH, Tsai CY. Post-acute care for frail older people decreases 90-day emergency room visits, readmissions and mortality: An interventional study. PLoS One. 2023 Jan 6;18(1):e0279654. doi: 10.1371/journal.pone.0279654. eCollection 2023. PMID 36607971